CLINICAL TRIAL: NCT06683560
Title: Evaluation of 3D Printed Aligners for Nasoalveolar Molding in Infants Born With Unilateral Complete Cleft Lip and Palate
Brief Title: Printed Aligners for Nasoalveolar Molding Treatment
Acronym: NAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maha Sabry Sayed, assistant lecturer, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Nasoalveolar molding
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Unilateral Complete Cleft Lip and Palate
Keywords: 3-dimensional; aligner; NAM; segmentation; Approximation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- infants born with complete unilateral cleft lip and palate (Experimental): photopolymer resin material "graphy" Tera Harz 85 will be used to print 3D printed aligners for nasoalveolar molding treatment
  Interventions: Device: : photopolymer resin material "graphy" Tera Harz 85 will be used to print 3D printed aligners for NAM treatment

INTERVENTIONS:
Device: : photopolymer resin material "graphy" Tera Harz 85 will be used to print 3D printed aligners for NAM treatment — 3d printed NAM aligner is made from novel photopolymer resin as a novel device
  Other Names: NAM device; NAM aligner

SUMMARY:
study will provide nasoalveolar molding (NAM) treatment, special care for infants born with cleft lip and palate. This novel appliance will help to provide the care in accurate and easy form by help of both digital work flow and new material which provide a unique properties.

DETAILED DESCRIPTION:
A sample of 10 infants born with unilateral cleft lip and palate (UCLP) ranging in age from seven to 45 days who meet the inclusion criteria will be recruited and subjected to the following study procedures: maxillary impression, extraoral scanning for nasolabial area and facial photos.

For digital workflow; the following steps will be done:

1. Digital model preparation.
2. Model segmentation and modification.
3. Virtual treatment simulation.
4. Virtual appliance construction.
5. Three-dimensional aligner printing.

After aligners printing, each infant will be delivered his own set of aligners. The nasal stent will be fixed to the aligner then delivered with a meticulous demonstration for parents regarding adhesive placement, insertion, and removal. Parents will be instructed to remove the aligner once per day for proper cleaning.

Infants will be followed up every two weeks till maxillary arch segments approximation and improvement of nasolabial tissue morphology. Finally, post-treatment records will be taken.

• Study Setting: The study will be performed in the clinic of the Orthodontic Department, Faculty of Dentistry, Ain-Shams University.

• Study procedure: Infants who meet the inclusion criteria and approve participation in the study will be included. An informed consent will be signed by the infant's parents before their enrollment in the study in which the aim of the study, the methodology, and possible complications will be clearly described. This research will be reviewed by the Research Ethics Committee, Faculty of Dentistry, Ain Shams University.

IX. Statistical Analysis Methods of assessment

1. Pre-operative T1 and postoperative T2 models will be digitally measured, assessed and compared.
2. Pre-operative T1 and postoperative T2 soft tissue scans will be digitally measured, assessed and compared.
3. Final virtual models and final infant models will be digitally compared.
4. Total treatment duration will be calculated. Finally, data will be tabulated and statistically analyzed

ELIGIBILITY:
Inclusion Criteria

1. Non-syndromic complete unilateral cleft lip, alveolus, and palate.
2. Age is up to 45 days.
3. Cleft size more than 5mm between anterior margins of cleft segments.

Exclusion Criteria

1. Infants are diagnosed with other congenital malformations.
2. Parents refusing NAM treatment.
3. Parents are unable to attend the clinic every 2 weeks.
4. Infants are born with another form of clefts like facial and median clefts.

Max Age: 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
approximation of segments of maxillary arch | almost 1.5 month
  measuring the alveolar cleft size before and after the treatment to assess the amount of cleft reduction on the scanned models in millimeter

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain shams univerisity, Cairo, Abbasya
  - Maha sabry Sayed, Cairo

IPD SHARING:
Plan to Share IPD: Yes
patients age, severity of malocclusion, photos
Supporting Information: Study Protocol
Time Frame: 11/2024 12/2025
Access Criteria: Noha Ibrahim google drive 11/2024

REFERENCES:
- [Background] Batra P, Raghavan S, Gribel BF. Nasoalveolar molding appliances. Am J Orthod Dentofacial Orthop. 2021 Feb;159(2):e85. doi: 10.1016/j.ajodo.2020.11.017. No abstract available. PMID 33546838